CLINICAL TRIAL: NCT05259072
Title: carDIo-ttranSSfOrm nucLEar Imaging Study
Acronym: DISSOLvE
Status: Terminated | Type: Observational
Why Stopped: Rolled over into another study
Sponsor: Oregon Health and Science University (Other)
Collaborators: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Ahmad Masri, Associate Professor, Oregon Health and Science University
Other Study IDs: 00023310
Record Dates: First submitted 2022-02-17; First posted 2022-02-28 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Amyloidosis; Transthyretin Amyloid Cardiomyopathy
Keywords: pyrophosphate scintigraphy; bone scintigraphy; eplontersen; tafamidis
MeSH Terms: conditions — Amyloidosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with transthyretin amyloid cardiomyopathy enrolled in CARDIO-TTRansform: Patients will undergo serial Tc-99m PYP imaging at baseline, week 61 and end of trial
  Interventions: Diagnostic Test: 99m-technetium pyrophosphate scintigraphy

INTERVENTIONS:
Diagnostic Test: 99m-technetium pyrophosphate scintigraphy — Imaging test
  Other Names: Tc-99m PYP

SUMMARY:
The investigators will evaluate the change in myocardial uptake of 99m-technetium pyrophosphate (Tc-99m PYP) tracer on serial planar and SPECT imaging in patients enrolled in the CARDIO-TTRansform clinical trial (NCT04136171).

DETAILED DESCRIPTION:
This is a multicenter trial of 80 subjects enrolled in the CARDIO-TTRansform randomized clinical trial (NCT04136171) who will undergo baseline and follow up Tc-99m PYP to assess for the change in myocardial uptake of the tracer.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were screened and eligible to be enrolled or have been already enrolled in the CARDIO-TTRansform randomized clinical trial (NCT04136171) and have a baseline 99m-technetium pyrophosphate planar and SPECT imaging done within 12 months prior to screening for CARDIO-TTRansform.
* Patients have to meet the inclusion and exclusion criteria of CARDIO-TTRansform trial to be enrolled.
* Patient willing to consent for the study and undergo the study procedures.

Exclusion Criteria:

* None

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ATTR-CM
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2022-01-19 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Primary outcome | 120-140 weeks
  Percentage of patients in both treatment groups with an improvement in the semi-quantitative visual grade by at least 1 grade from baseline and an improvement in the heart/contralateral ratio by at least 20% from baseline to end of treatment.

SECONDARY OUTCOMES:
Secondary outcome | 120-140 weeks
  Change in cardiac amyloid activity on Tc-99m PYP SPECT as quantified by the target to background ratio from baseline to end of treatment
Secondary outcome | 61 weeks
  Percentage of patients in both treatment groups with an improvement in the semi-quantitative visual grade by at least 1 grade from baseline and an improvement in the heart/contralateral ratio by at least 20% from baseline to week 61

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Masri, MD MS, Study Chair — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No